CLINICAL TRIAL: NCT00929253
Title: Efficacy of Computer Delivered CRA (Bup II) Grant No. R01DA012997-10
Brief Title: Efficacy of Computer Delivered Community Reinforcement Approach (CRA) (Bup II)
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Warren K. Bickel, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 31695
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Opiate Addiction
Keywords: Opioid Dependence; Opiates; Hydrocodone; Oxycodone; Oxycontin; Narcotic Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer delivered CRA + CM + Suboxone (Active Comparator): In this arm, participants are administered Suboxone and therapy is delivered by a computer. Fluency training is provided. The participant then listens through headphones and reads the information on the screen. They progress through various modules that involve education regarding high risk situations for potential use drug and skills to deal with those situations. In addition, skills for dealing with anxiety and anger are also provided. Videos are displayed that have examples of real-left situations. HIV/AIDS education is also provided. The program is interactive with the participant being required to answer short questions at the end of each module and prompts for "homework" worksheets are provided. These participants receive vouchers for providing drug negative urine samples.
  Interventions: Drug: Suboxone; Behavioral: CRA; Behavioral: Therapy; Behavioral: CM
- CM + Suboxone (Active Comparator): In this arm of the study, the participants receive vouchers for providing a drug negative urine sample. These participants, however, do not have computer delivered therapy.
  Interventions: Drug: Suboxone; Behavioral: Therapy; Behavioral: CM

INTERVENTIONS:
Drug: Suboxone — Dosage Form: Oral Tablet; Dosage 6, 12, or 18 mg; Frequency; Daily; Duration 12 weeks
  Other Names: Buprenorphine
Behavioral: CRA — Computer-delivered Community Reinforcement Approach
  Arms: Computer delivered CRA + CM + Suboxone
Behavioral: Therapy — Therapist-delivered therapy
Behavioral: CM — Contingency management (vouchers) for providing a drug negative urine sample.

SUMMARY:
This study is designed to examine the effects of combined buprenorphine and voucher incentives to promote abstinence from illicit opiate use, along with or without computer-delivered therapy, during treatment of opioid dependence.

DETAILED DESCRIPTION:
The Community Reinforcement Approach (CRA) with contingency management (CM) is a widely researched and demonstrably efficacious drug abuse treatment. This treatment is derived from drug self-administration research and a behavioral analysis of drug dependence, where abused drugs are thought to compete successfully with the more delayed pro-social reinforcers because of their relatively more immediate reinforcing effects. The CRA treatment with CM approach takes this theoretical view into account by (1) providing immediate positive reinforcement for abstinence via the voucher reinforcement procedure, and (2) having therapists teach skills and encourage behaviors that help improve employment status, family/social relations and increase recreational activities via the CRA treatment. The incentives for abstinence with the enhancement of non-drug sources of reinforcement are then expected to successfully compete with the reinforcement from drug use. Adoption of CRA with CM may be facilitated if it could be delivered so that it is both less costly and requires less staff time to implement. In our previous trial, we demonstrated that among buprenorphine maintained opioid-dependent persons, computer-delivered CRA with CM (i.e., voucher incentives) was as effective as and less costly than therapist-delivered CRA with CM (i.e., voucher incentives). However, the design of that study did not indicate whether the computer-delivered CRA produced increases in abstinence over that produced by the CM (i.e., voucher incentives) procedures alone. Thus, we believe the contribution of the computerized treatment to therapeutic outcomes should be isolated.

In this study, which will include only buprenorphine maintained opioid-dependent participants, we plan to examine whether computer-delivered CRA produces increases in abstinence over that produced by CM (i.e., voucher incentives) procedures alone. Specifically, this trial will compare computer-delivered CRA with vouchers (with minimal therapist involvement) and voucher incentives alone in a randomized parallel groups design. Participants will be assigned randomly to receive one of two treatments: (1) computer-delivered CRA along with voucher incentives (i.e., CM); or (2) voucher incentives (i.e., CM) alone. Outcome measures will include abstinence and retention. We hypothesize that the computer-delivered CRA with CM will be more efficacious than CM.

Importantly, in this trial, the treatment interventions will reinforce both cocaine and opioid abstinence. Many opioid-dependent individuals also abuse, or are dependent upon, cocaine and polydrug abuse in this population has been rarely addressed. By targeting both drugs, our understanding of effective ways to address polydrug abuse will be increased.

Overall, this research will contribute new empirical information regarding the efficacy of providing CRA with CM. Such information may result in more cost-effective treatment and facilitate its dissemination. This research will further examine the utility of computerizing a substantive portion of substance abuse treatment. Computerization of treatment is a novel approach that may positively impact the future of drug abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* history of opioid dependence
* significant current opioid use

Exclusion Criteria:

* unstable medical or psychiatric conditions
* pregnancy
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2007-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, Ph.D., Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bickel WK, Marsch LA, Buchhalter AR, Badger GJ. Computerized behavior therapy for opioid-dependent outpatients: a randomized controlled trial. Exp Clin Psychopharmacol. 2008 Apr;16(2):132-43. doi: 10.1037/1064-1297.16.2.132. PMID 18489017
- [Result] Kirshenbaum AP, Olsen DM, Bickel WK. A quantitative review of the ubiquitous relapse curve. J Subst Abuse Treat. 2009 Jan;36(1):8-17. doi: 10.1016/j.jsat.2008.04.001. Epub 2008 Jun 24. PMID 18571890
- [Derived] Maricich YA, Bickel WK, Marsch LA, Gatchalian K, Botbyl J, Luderer HF. Safety and efficacy of a prescription digital therapeutic as an adjunct to buprenorphine for treatment of opioid use disorder. Curr Med Res Opin. 2021 Feb;37(2):167-173. doi: 10.1080/03007995.2020.1846022. Epub 2020 Dec 7. PMID 33140994
- [Derived] Christensen DR, Landes RD, Jackson L, Marsch LA, Mancino MJ, Chopra MP, Bickel WK. Adding an Internet-delivered treatment to an efficacious treatment package for opioid dependence. J Consult Clin Psychol. 2014 Dec;82(6):964-72. doi: 10.1037/a0037496. Epub 2014 Aug 4. PMID 25090043
- See also: Click here to learn more about drug addiction studies at the Fralin Biomedical Research Institute at Virginia Tech Carilion — https://fbri.vtc.vt.edu/people-directory/primary-faculty/bickel.html

RESULTS

PARTICIPANT FLOW:
Groups:
- CM + Suboxone: In this arm of the study, the participants receive vouchers for providing a drug negative urine sample. These participants, however, do not have computer delivered CRA, only treatment as usual with a biweekly 30-minute meeting with a clinician.
  Suboxone: Dosage Form: Oral Tablet; Dosage 6, 12, or 18 mg; Frequency; Daily; Duration 12 weeks
  Therapy: treatment as usual
  CM: Contingency management (vouchers) for providing drug negative urine samples.
Period: Overall Study
Arm/Group | Computer Delivered CRA + CM + Suboxone | CM + Suboxone
Started | 91 | 79
Completed | 91 | 79
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CM + Suboxone: In this arm of the study, the participants receive vouchers for providing a drug negative urine sample. These participants, however, do not have computer deliver therapy, only treatment as usual consisting of biweekly 30-minute counseling sessions.
  Suboxone: Dosage Form: Oral Tablet; Dosage 6, 12, or 18 mg; Frequency; Daily; Duration 12 weeks
  Therapy: treatment as usual
  CM: Contingency management (vouchers) for providing a drug negative urine sample.
- Total: Total of all reporting groups
Arm/Group | Computer Delivered CRA + CM + Suboxone | CM + Suboxone | Total
Number analyzed (Participants) | 91 | 79 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.85) | 33.6 (9.8) | 32.9 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 32 | 78
  Male | 45 | 47 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 91 | 79 | 170
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 87 | 75 | 162
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 91 | 79 | 170

OUTCOME MEASURES:

1. Primary Outcome: Abstinence
Description: Abstinence defined as the longest documented period of continuous abstinence from opioids and cocaine
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Groups:
- CM + Suboxone: In this arm of the study, the participants receive vouchers for providing a drug negative urine sample. These participants, however, do not have computer deliver therapy.
  Suboxone: Dosage Form: Oral Tablet; Dosage 6, 12, or 18 mg; Frequency; Daily; Duration 12 weeks
  Therapy: Therapist-delivered therapy
  CM: Contingency management (vouchers) for providing a drug negative urine sample.
Arm/Group | Computer Delivered CRA + CM + Suboxone | CM + Suboxone
Number analyzed (Participants) | 91 | 79
days | 55.0 (26.2) | 49.5 (30.6)

ADVERSE EVENTS:
Description: Adverse event data were collected throughout the clinical trial from 2007 to 2010. At the time of the conduct of the clinical trial, adverse events were monitored by specific type. At this time (over ten years after data collection and five years after publication of the data), specific details are not available.
Arm/Group | Computer Delivered CRA + CM + Suboxone | CM + Suboxone
Serious Adverse Events (participants affected / at risk) | 0/91 | 0/79
Other Adverse Events (participants affected / at risk) | 57/91 | 55/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Computer Delivered CRA + CM + Suboxone (N=91) | CM + Suboxone (N=79)
adverse event (General disorders) | 57 (147) | 55 (113)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No